CLINICAL TRIAL: NCT00331669
Title: Multicenter, Randomized Trial on the Effects of Pallidal Deep Brain Stimulation for Tardive Dystonia
Brief Title: Efficacy and Safety of Deep Brain Stimulation (DBS) of the Pallidal (GPi) in Patients With Tardive Dystonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Humboldt-Universität zu Berlin (Other); Ruhr University of Bochum (Other); Medical University of Cologne (Other); Heinrich-Heine University, Duesseldorf (Other); University Hospital Freiburg (Other); Medical University of Hannover (Other); Medical University Innsbruck (Other); University of Kiel (Other); Philipps University Marburg (Other); Ludwig-Maximilians - University of Munich (Other); University of Rostock (Other); University of Regensburg (Other); University Hospital Tuebingen (Other); Medical University of Vienna (Other); Medtronic (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DBS and tardive dystonia
Record Dates: First submitted 2006-05-26; First posted 2006-05-31 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-02

CONDITIONS: Dystonia; Movement Disorder
Keywords: deep brain stimulation; pallidum; tardive dystonia; randomized; double blind; multicenter
MeSH Terms: conditions — Dystonia; Movement Disorders; Tardive Dyskinesia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Placebo Comparator): device
  Interventions: Procedure: deep brain stimulation

INTERVENTIONS:
Procedure: deep brain stimulation — high frequency stimulation

SUMMARY:
The purpose of this randomized, double blind, multi-center study is to assess the efficacy and safety of bilateral pallidal deep brain stimulation in patients with tardive dystonia.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) has been established as a new reversible, neurosurgical therapeutic option for patients suffering from disabling neurological movement disorders such as essential tremor and Parkinson´s disease. Recently, deep brain stimulation has been successfully applied in patients with primary generalized and segmental dystonia. Additionally, a number of case reports suggest that pallidal deep brain stimulation may also improve tardive dystonia, which may for instance result from the intake of neuroleptics and which is notoriously difficult to treat medically. The present study will investigate the effects of pallidal DBS using a double blind, randomized design (sham- versus verum-stimulation within a 3-months interval post implantation of the electrodes).

Initially 60 patients had been calculated in a power analysis to assess significant results based on an average improvement of dystonic symptoms of 30%. However, in a recent study (Damier et al., Archives of General Psychiatry, 2007), 10 out of 10 showed a successful outcome of approximately 50% decrease on the extrapyramidal symptoms rating scale score. The exact one- sided lower 95% confidence limit would be 0.794 for this result. If such an approach is chosen for sample size estimation with 18 verum and 18 placebo patients one would obtain a power of 82% against a placebo effect of 30% success rate. For a placebo effect of 25% one needs 16+16 patients and for the placebo effect of 20% one needs 12+12 patients. We thus decided to reduce the sample size to 36- 32- 24 patients. It is expected that the continuous primary outcome measure will preserve even higher power than the binary one used in the study mentioned above. The local ethical committee has approved this.

ELIGIBILITY:
Inclusion Criteria:

* Operational criteria for tardive dystonia for > 18 months after cessation of neuroleptic exposure
* 18-75 years
* Relevant functional impairment in daily living activities
* BFMDRS > 8 or AIMS > 16
* Informed written consent

Exclusion Criteria:

* PANNS >60 (Schizophrenia)
* Hamilton-Score > 18 (Depression)
* MATTIS-Score <120 (Dementia)
* Preceding stereotactic neurosurgery
* Pronounced brain atrophy
* Increased bleeding risk
* Decreased immune status
* Botulinum Toxin treatment within the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-05; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of the motor scale of Burke-Fahn-Marsden-Dystonia Rating Scale via blinded video assessment 3 months after starting DBS in comparison to sham-stimulated patients | 3 months

SECONDARY OUTCOMES:
AIMS | 3 months
Non-motor subscores of BMFDRS | 3 months
Visual analogue scales for both patients and treating physicians | 3 months
Quality of life (SF-36) | 3 months
Psychiatric assessment (HADS-D and PANSS) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas R Kupsch, MD, Principal Investigator — Dpt. of Neurology, Augustenburger Platz 1, 13353 Berlin, Charite, Campus Virchow, Germany
Locations (1):
- Andreas Kupsch, Berlin, Germany

REFERENCES:
- [Background] Trottenberg T, Volkmann J, Deuschl G, Kuhn AA, Schneider GH, Muller J, Alesch F, Kupsch A. Treatment of severe tardive dystonia with pallidal deep brain stimulation. Neurology. 2005 Jan 25;64(2):344-6. doi: 10.1212/01.WNL.0000149762.80932.55. PMID 15668437
- [Background] Franzini A, Marras C, Ferroli P, Zorzi G, Bugiani O, Romito L, Broggi G. Long-term high-frequency bilateral pallidal stimulation for neuroleptic-induced tardive dystonia. Report of two cases. J Neurosurg. 2005 Apr;102(4):721-5. doi: 10.3171/jns.2005.102.4.0721. PMID 15871516
- [Background] Damier P, Thobois S, Witjas T, Cuny E, Derost P, Raoul S, Mertens P, Peragut JC, Lemaire JJ, Burbaud P, Nguyen JM, Llorca PM, Rascol O; French Stimulation for Tardive Dyskinesia (STARDYS) Study Group. Bilateral deep brain stimulation of the globus pallidus to treat tardive dyskinesia. Arch Gen Psychiatry. 2007 Feb;64(2):170-6. doi: 10.1001/archpsyc.64.2.170. PMID 17283284
- [Derived] Gruber D, Sudmeyer M, Deuschl G, Falk D, Krauss JK, Mueller J, Muller JU, Poewe W, Schneider GH, Schrader C, Vesper J, Volkmann J, Winter C, Kupsch A, Schnitzler A; DBS study group for dystonia. Neurostimulation in tardive dystonia/dyskinesia: A delayed start, sham stimulation-controlled randomized trial. Brain Stimul. 2018 Nov-Dec;11(6):1368-1377. doi: 10.1016/j.brs.2018.08.006. Epub 2018 Sep 11. PMID 30249417